CLINICAL TRIAL: NCT00999037
Title: FGF-23 (Fibroblast Growth Factor 23) Regulation in Chronic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1K23DK080984-01A1 (NIH)
Record Dates: First submitted 2009-10-20; First posted 2009-10-21 (Estimated); Results first posted 2017-03-31 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Secondary Hyperparathyroidism
MeSH Terms: conditions — Hyperparathyroidism, Secondary | interventions — Sevelamer

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Renvela (Experimental): Daily renvela with meals for 12 weeks
  Interventions: Drug: Sevelamer Carbonate
- placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Sevelamer Carbonate — Daily renvela (800 mg tid with meals) x 12 weeks
  Other Names: Renvela
  Arms: Renvela
Other: Placebo — 1 inert tablet tid x 12 weeks
  Arms: placebo

SUMMARY:
FGF-23 is a newly described protein that is an important regulator of phosphorus in the body. This protein increases in people with kidney disease and people who need dialysis have very high levels of FGF-23 in the blood. However, although some studies have indicated that FGF-23 levels go up with increased intake of phosphorus, no one knows if FGF-23 levels can be lowered in patients with kidney disease by preventing them from absorbing phosphorus from food. This study is designed to see what happens to levels of FGF-23 in the blood when patients with chronic kidney disease take medications to prevent phosphorus absorption. Since high levels of FGF-23 have been linked with increased rates of death in patients with advanced kidney disease, controlling the levels may, in the future, be a way to decrease heart disease in patients with kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria include pediatric patients, between the ages of 2 and 21 years, with CKD stages 2-4 (GFR 15-90 ml/min/1.73m2).

Exclusion Criteria:

* Exclusion criteria include: the use of phosphate binder therapy within the past 3 months, treatment with 25(OH)vitamin D or 1,25dihydroxyvitamin D, underlying metabolic bone disease, or underlying renal phosphate wasting disorder.

Ages: 6 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2009-10; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Renvela: Sevelamer Carbonate (Renvela) 800 mg tablets: 1 tablet TID with meals for 12 weeks
- Placebo: Placebo (inert tablets): 1 tablet TID with meals for 12 weeks
Period: Overall Study
Arm/Group | Renvela | Placebo
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Renvela | Placebo | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9 | 6 | 15
  Between 18 and 65 years | 0 | 3 | 3
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.3 (3.2) | 15.4 (4.6) | 14.3 (4.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 4 | 5 | 9
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Change in FGF-23 Level
Description: Change in FGF23 value from baseline in response to Renvela at 12 weeks in comparison to placebo.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Groups:
- Renvela: Sevelamer Carbonate (800 mg tablet) PO TID with meals x 12 weeks
- Placebo: Placebo (1 inert tablet) PO TID with meals x 12 weeks
Arm/Group | Renvela | Placebo
Number analyzed (Participants) | 9 | 9
percentage change from baseline | 16 (41) | 41 (46)

2. Secondary Outcome: 1,25(OH)2vitamin D Value
Description: Percentage change in 1,25(OH)2vitamin D level from baseline at 12 weeks.
Time Frame: 12 week
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Renvela | Placebo
Number analyzed (Participants) | 9 | 9
percent change from baseline | 82 (64) | 69 (82)

3. Secondary Outcome: Serum Phosphate Concentration
Description: Change in serum phosphate at 12 weeks from baseline
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Renvela | Placebo
Number analyzed (Participants) | 9 | 9
percent change from baseline | -4 (46) | -8 (49)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Renvela | Placebo
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No